CLINICAL TRIAL: NCT02183714
Title: The Ability of Songha Night ® to Improve Sleep in Patients With Mild to Moderate Sleep Disturbances
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 582.1
Record Dates: First submitted 2014-07-07; First posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Sleep Initiation and Maintenance Disorders
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

ARMS (2):
- Songha Night ® (Experimental)
  Interventions: Drug: Songha Night ®
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Songha Night ®
  Arms: Songha Night ®
Drug: Placebo
  Arms: Placebo

SUMMARY:
To evaluate the effect of Songha Night ® on insomnia, anxiety and quality of life compared to placebo in patients with mild to moderate insomnia.

ELIGIBILITY:
Inclusion Criteria:

* Psychophysiologic insomnia
* Severity: mild to moderate
* Duration: subacute to chronic
* Subjects age > 18 and < 65, men or women
* Subject had to give written informed consent

Exclusion Criteria:

* Regular use of psycho-active drugs
* Work in shifts
* Use of psychoactive drugs during the past 30 days
* Any treatment that might interfere with his/her participation in this study and the evaluation of the efficacy or safety of the test drug (e.g. renal insufficiency, hepatic or metabolic dysfunction, cardiovascular disease, psychiatric disorder, myasthenia gravis, delirious state, etc.)
* known hypersensitivity to any of the ingredients of the study drug
* Pregnancy, lactation, women of childbearing potential not using an established contraceptive
* Drug and alcohol abuse
* Participation in another trial within the past 30 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 1998-05; Primary Completion 1998-12 (Actual)

PRIMARY OUTCOMES:
Change in sleep quality on a 100 mm visual analogue scale (VAS) | baseline, after 2 and 4 weeks of treatment, 1 week after end of treatment

SECONDARY OUTCOMES:
Feeling refreshed score (six point rating scale) | up to week 5
Ability to concentrate and perform well score (six point rating scale) | up to week 5
Night-time total sleeping time | up to week 5
Difficulty in falling asleep (five point rating scale) | up to week 5
Number of awakenings during the night | up to week 5
Physical and mental health state by short form (SF-36) questionnaire | up to week 5
Anxiety by State-Trait Anxiety Inventory | up to week 5
Frequency of adverse events | up to week 5
Global clinical impression on insomnia by short questionnaire | up to week 5